CLINICAL TRIAL: NCT05665829
Title: Randomised Controlled Trial of Awake Transnasal Laser-assisted Surgery (TNLS) and Microlaryngeal Surgery for Benign Laryngeal Lesions
Brief Title: Awake Transnasal Laser-assisted Surgery (TNLS) and Microlaryngeal Surgery for Benign Laryngeal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tam Aurora Ka Yue, Clinical Tutor (honorary), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CREC Ref. No. 2021.170
Record Dates: First submitted 2022-12-06; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Awake Laser; Microlaryngeal Surgery; Benign Laryngeal Lesion; Transnasal Laser Surgery

STUDY DESIGN:
Intervention Model Description: This is a prospective randomised controlled trial
Masking Description: non
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microlaryngeal surgery (MLS) (Active Comparator): For traditional MLS under general anesthesia, after intubation with microlaryngeal tube, a laryngoscope will be inserted transorally under direct vision and suspended. Laryngeal lesions are visualized with either microscope or endoscope, and removed with microsurgery instruments and sent for routine section
  Interventions: Procedure: Microlaryngeal surgery (MLS)
- Awake transnasal laser-assisted surgery (TNLS) (Experimental): For TNLS, a transnasal channel flexible laryngoscope is used with prior trans-nasal, trans-oral and trans-laryngeal local anesthesia application. A 445nm blue laser is introduced via a working channel of laryngoscope, with a lesion-specific laser setting. Biopsy can be performed by devascularizing and thinning the lesion down to a pedicle, then removed with biopsy forcep. During the operation, patient will receive continuous SpO2 monitoring with regular blood pressure monitoring. Patients are discharged on same day of procedure after close observation for 2 hours in day center.
  Interventions: Procedure: Awake transnasal laser-assisted surgery (TNLS)

INTERVENTIONS:
Procedure: Awake transnasal laser-assisted surgery (TNLS) — The experimental intervention would be awake transnasal laser-assisted surgery under local anesthesia, carried out in minor operation theater as a day-case basis in ENT ambulatory center.
  Arms: Awake transnasal laser-assisted surgery (TNLS)
Procedure: Microlaryngeal surgery (MLS) — For traditional MLS under general anesthesia, laryngeal lesions are visualized and removed with under microscopic or endoscopic approach.
  Arms: Microlaryngeal surgery (MLS)

SUMMARY:
This is a prospective, single-cluster randomised controlled trial conducted at two tertiary referral hospitals in Hong Kong to compare the clinical and functional outcomes of office-based transnasal laser-assisted surgery (TNLS) under local anesthesia to traditional microlaryngeal surgery (MLS) under general anesthesia.

DETAILED DESCRIPTION:
Patients with benign laryngeal lesions were block-randomized to either TNLS or traditional MLS group. Pre-operative diagnosis and post-operative follow-up were conducted in a multidisciplinary voice clinic. All patients were followed up at 2-week, 6-week, 3-month, 6-month and 1-year post-operation. Primary outcome included functional vocal measures using Voice-Handicap index (VHI-30). Secondary outcomes included length of stay, patient-perceived procedural discomfort, complications, operative time, recurrence rate, reoperation rate, and medical cost.

ELIGIBILITY:
Inclusion Criteria:

* older than 18-year-old
* mentally competent to give an informed consent
* operable benign laryngeal lesions
* able to tolerate transnasal flexible laryngoscopy

Exclusion Criteria:

* under 18-year old
* unable to give an informed consent
* unable to tolerate flexible laryngoscopy under local anesthesia
* allergy to local anesthesia
* unfavourable anatomy precluding adequate visualization
* with extensive lesions with expected difficult operation
* with pathologies suspicious of or confirmed malignancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Voice-Handicap Index (VHI-30) | Post-op 2 week
  The VHI-30 is a 30-item self-administered questionnaire, which is a reliable measure for voice treatment outcome.It consists of three subscales, namely physical, functional and emotional. It provides an overall measurement of a person's vocal function and how it influences on a person's everyday functioning and experience. It has a overall score range from 0 to 120, 0 as the best score, 120 as the worst score.
Voice-Handicap Index (VHI-30) | Post-op 6 week
  The VHI-30 is a 30-item self-administered questionnaire, which is a reliable measure for voice treatment outcome.It consists of three subscales, namely physical, functional and emotional. It provides an overall measurement of a person's vocal function and how it influences on a person's everyday functioning and experience. It has a overall score range from 0 to 120, 0 as the best score, 120 as the worst score.
Voice-Handicap Index (VHI-30) | Post-op 3 month
  The VHI-30 is a 30-item self-administered questionnaire, which is a reliable measure for voice treatment outcome.It consists of three subscales, namely physical, functional and emotional. It provides an overall measurement of a person's vocal function and how it influences on a person's everyday functioning and experience. It has a overall score range from 0 to 120, 0 as the best score, 120 as the worst score.
Voice-Handicap Index (VHI-30) | Post-op 6 month
  The VHI-30 is a 30-item self-administered questionnaire, which is a reliable measure for voice treatment outcome.It consists of three subscales, namely physical, functional and emotional. It provides an overall measurement of a person's vocal function and how it influences on a person's everyday functioning and experience. It has a overall score range from 0 to 120, 0 as the best score, 120 as the worst score.
Voice-Handicap Index (VHI-30) | Post-op 1 year
  The VHI-30 is a 30-item self-administered questionnaire, which is a reliable measure for voice treatment outcome.It consists of three subscales, namely physical, functional and emotional. It provides an overall measurement of a person's vocal function and how it influences on a person's everyday functioning and experience. It has a overall score range from 0 to 120, 0 as the best score, 120 as the worst score.

SECONDARY OUTCOMES:
Procedure-oriented outcomes | Intraoperative
  Operation time
Procedure-oriented outcomes | Intraoperative
  Completeness of lesion removal
Procedure-oriented outcomes | Intraoperative
  Complications in Clavien-Dindo classification
Procedure-oriented outcomes | Perioperative
  Length of hospital stay
Procedure-oriented outcomes | Post-op 2 week, 6 week, 3 month, 6 month, 1 year
  Recurrence rate
Procedure-oriented outcomes | 1 year
  Reoperation
Cost | Peri-operative
  Medical costs including surgery-related and hospitalization-related costs are estimated.
Patient-perceived procedural discomfort | Immediate post-operation
  Discomfort in visual analog scale, from 0 to 10, 0 as least discomfort, 10 as most uncomfortable.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong